CLINICAL TRIAL: NCT00592319
Title: Voice-preserving Treatment of Laryngeal Papilloma
Brief Title: Celebrex (Celecoxib) Treatment of Laryngeal Papilloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: 03/01/2009,due to date close to termination of this funding/study period
Sponsor: Boston University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Zhi Wang, Professor and Director, Boston University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDC-006617A; R01DC006617 (NIH)
Record Dates: First submitted 2007-12-31; First posted 2008-01-14 (Estimated); Results first posted 2012-08-24 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Laryngeal Papilloma
Keywords: Papilloma; pulsed dye laser; Celebrex; voice
MeSH Terms: conditions — Laryngeal papillomatosis; Papilloma | interventions — Celecoxib; Lasers, Gas; Microsurgery; Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PDL+Celebrex (Experimental): endoscopic treatment with once-time PDL radiation at 6.0-8.0 J on laryngeal papilloma, followed by oral taking of 9-month Celebrex (100mg, BID), in 15 subjects
  Interventions: Drug: Celebrex; Device: PDL
- standard surgery (Active Comparator): once-time and routine surgery, with either of carbon dioxide (CO2) laser radiation at 10.0-20.0 W or "cold" surgery with microinstruments, in 15 subjects
  Interventions: Procedure: CO2 laser or microsurgery

INTERVENTIONS:
Drug: Celebrex — oral taking of Celebrex (100 mg, BID) for 9 months
  Other Names: Celecoxib
  Arms: PDL+Celebrex
Device: PDL — once time radiation on laryngeal papilloma with PDL , at 6.0-8.0 J
  Other Names: 585 nm PDL (cynosure Inc. Mass)
  Arms: PDL+Celebrex
Procedure: CO2 laser or microsurgery — once-time surgery to remove laryngeal papilloma
  Other Names: ablation laser or micro-instrumental surgery
  Arms: standard surgery

SUMMARY:
Respiratory recurrent papilloma (RRP) is one of the most common benign tumors. Surgical removal is the current management for RRP, but it is a very traumatic procedure, and often leads to permanent voice dysfunction. In this study, we will develop a new, combined RRP treatment with a pulsed dye laser (PDL) and Celebrex. We will determine if Celebrex, a newly developed inhibitor of cyclooxygenase (COX)-2, can provide a long-term inhibitory effect on RRP, therefore preventing RRP from recurring. This combined strategy, if successful in this proposed study, will provide a new and ideal "voice-preserving" therapy for RRP that will deliver long-term efficacy in managing RRP.

DETAILED DESCRIPTION:
RRP and its surgeries usually involves the vocal cords or other regions of the larynx, thereby, resulting in a poor voice. Our previous studies have shown the efficacy and safety of a microvascular targeting technique (MVT) for RRP treatment using the 585 nm PDL. This technique provides a less traumatic alternative to surgery. However, postoperative recurrence of lesions still remains a problem because of microvascular regrowth. This study is a continuation of our effort to develop a new and less traumatic treatment for RRP. In this study, we will develop a new, combined RRP treatment with PDL and Celebrex. We will determine if Celebrex, a newly developed inhibitor of COX-2, can provide a long-term inhibitory effect on RRP through its anti-angiogenic activity and the synergic effect produced with the laser therapy. The hypothesis is that postoperative administration of Celebrex will provide a long-term inhibitory effect on microvascular regrowth and on COX-2 enzyme, thereby, preventing RRP from recurring after the PDL therapy. Our specific aim in this study is to determine the synergic effect between PDL and Celebrex and long-term efficacy of Celecoxib in preventing postoperative RRP recurrence. We will compare this new combined strategy with traditional treatments in 30 adult patients. This is the first time to combined this new laser MVT technique with a COX-2 inhibitor for microvascular targeting therapy of RRP. This combined strategy, if successful in this proposed study, will provide a new and ideal "voice-preserving" therapy for RRP that will deliver long-term efficacy in managing RRP and will be safe and convenient enough for use in out-patient treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 64 years of age
2. with laryngeal papillomas requiring surgical treatment
3. willingness to participate in the study
4. a signed informed consent form

Exclusion Criteria:

1. age less than 18 years
2. evidence of mental impairment so that the patient can not understand or sign the consent form
3. malignant diseases such as laryngeal cancer
4. established coronary heart and artery disorder, cerebrovascular disease, and other cardiovascular diseases
5. established diabetes, which requires (1) insulin treatment; or (2) more than 2 oral agents of medication; or (3) to have a baseline HgbA1c >8.0
6. hypertension, with ongoing blood pressure > 150 mg Hg systolic or to require medication
7. family history with serious cardiovascular events and problems
8. any sign and evidence which in the opinion of cardiovascular physician warrants exclusion of subject

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2005-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wang Zhi, M.D, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 years
Pre-assignment Details: Many patients, who were eligible for this study, finally declined to participate this study due to a safety concern with Celebrex
Groups:
- Control: once-time routine surgery with (either of CO2 laser at continue model and 10.0-20.0 W, or "cold" surgery with micro-instruments), in 15 subjects
- Experimental: once-time PDL surgery at 6.0-8.0 W, followed by oral taking of Celecoxib (100mg,BID)for 9 months
Period: Overall Study
Arm/Group | Control | Experimental
Started | 2 | 8
Completed | 2 | 5
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Control: treated with routine surgery (CO2 laser or "cold" microsurgery), in 15 cases
- Experimental: treated with once-time PDL, followed by oral taking of 9-month Celecoxib, in 15 cases
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 2 | 8 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 8 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 1 | 4 | 5

OUTCOME MEASURES:

1. Secondary Outcome: Time Course (Month) With Papilloma Recurrence During 12-month Follow up
Description: The measuer is reported as time course (i.e., how many month) to see papilloma recurrence if there is any such recurrence.
Time Frame: 12 months
Population: 12-month follow-up
Measure: Mean (Full Range); unit: month
Groups:
- Control: treated with once-time routine surgery
- Experiment: treated with both of once-time PDL and 9-month Celebrex
Arm/Group | Control | Experiment
Number analyzed (Participants) | 2 | 5
month | 3.5 [3 to 4] | 5.2 [2 to 10]

2. Primary Outcome: Number of Case With Papilloma Recurrence During a 12-month Follow up
Description: Criteria for the recurrence: the site scoring >4, plus visible lesion found in >50% of the treated tissue area, after surgery Description: The caculation of the site scoring is based on a called Derkay's scoring system: to indicate how many anatomic site involved, from the 0 (the best)to 13 (the worst),among a total of 13 laryngeal sites such as epiglottis or right true vocal cords.
Time Frame: 12-month follow up
Population: The paticipants for analysis were those who had the recurrence or completed follow-up period. The analysis was per protocol, and follow-up period was 12 months.
Measure: Number; unit: case
Groups:
- Control: treated with once-time routine surgery (CO2 laser or "cold" microsurgery)
- Experienment: treated with once-time PDL, followed by oral taking of Celebrex (100mg,BID) for 9 months
Arm/Group | Control | Experienment
Number analyzed (Participants) | 2 | 5
case | 2 [0 to 0] | 5 [0 to 0]

ADVERSE EVENTS:
Time Frame: Primary: cardiovascular events for 12 months
Description: Others: laser and surgery complications for 12 months
Groups:
- Experiment: treated with both of PDL and Celecoxib
- Control: treatd with CO2 laser or microsurgery
Arm/Group | Experiment | Control
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/2
Other Adverse Events (participants affected / at risk) | 0/8 | 0/2

LIMITATIONS AND CAVEATS:
We failed to recruit a total of 30 cases, due to (1) This disease is relative less common in clinic; and (2) particularly, more and more of patients now had a serious concern in safety of Celebrex due to news and warnings to public in recent years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No